CLINICAL TRIAL: NCT04136834
Title: A Phase I Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Activity o f Ascending Doses of PT0I (Pegtomarginase) in Subjects With Advanced Malignancies
Brief Title: A Phase I Open-label Study for Subjects With Advanced Malignancies
Acronym: PT01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-PT01-001
Record Dates: First submitted 2019-10-01; First posted 2019-10-23 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegtomarginase (PT01) (Experimental): To determine the MTD of PT01 based on the toxicity observed during Cycle 1 of the Dose Escalation Phase and to investigate the safety and tolerability of PT01 when administered intravenously(IV) to subjects with advanced malignancies
  Interventions: Biological: PT01 (Pegtomarginase)

INTERVENTIONS:
Biological: PT01 (Pegtomarginase) — PT01 (Pegtomarginase) breaks down arginine in the blood stream, reducing the supply of arginine and stopping the cancer cells from growing. Normal cells can continue to make their own arginine inside the cell, so PT01 targets the rapidly growing cancer cells.

SUMMARY:
This is a first-in-human (FIH) Phase 1 dose escalation study to evaluate the safety, tolerability, PK, PD, and preliminary activity of PT01 administered IV in subjects with advanced malignancies.'

DETAILED DESCRIPTION:
The study consists of a Dose Escalation Phase and a Dose Expansion Phase, both of which include a 28-day Screening Period, Baseline, a Treatment Period (comprised of 28-day cycles with weekly dosing on Days 1, 8, 15, and 22), and a Follow-up Period. Unique to the Dose Escalation Phase is the inclusion of Cycle 0 during which a single dose of PT01 will be administered before Cycle 1 for detailed exploration of the PK/PD relationship.

All PT01 IV doses will be administered at the clinical site.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must have/be:

1. Able to understand and voluntarily sign an informed consent form (ICF)
2. Male and female adults ≥18 years of age at the time of informed consent
3. Advanced solid malignancies for which no standard therapy is available. Subjects in whom available standard therapy is contraindicated may be eligible.
4. For Dose Expansion Phase:

   • Expansion Group A: Histologically confirmed unresectable locally advanced or metastatic (AJCC stage IIIB, IIIC, or IV) cutaneous malignant melanoma for which no standard therapy is suitable.
5. At least 1 measurable site of disease as defined per RECIST v1.1 criteria (Dose Expansion Phase) or evaluable disease (Dose Escalation Phase only)
6. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
7. Life expectancy of >12 weeks
8. Adequate hematologic status within 28 days prior to dosing as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain:

   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Platelet count ≥100 × 109/L
   * Hemoglobin ≥90 g/L
9. Adequate liver function as demonstrated by:

   * Serum bilirubin <2 × the upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤3 × ULN or ≤5 × ULN in subjects with liver metastases
   * Gamma-glutamyl transferase ≤5 × ULN Athenex, Inc. Confidential Page 9 Final v2.0_17 Jun 2019 Clinical Study Protocol_Amendment 01 ATX-PT01-001
   * Alkaline phosphatase ≤3 × ULN or ≤5 × ULN if bone or liver metastasis is present
10. Serum creatinine ≤1.5 × ULN or estimated creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula
11. Prothrombin time(PT) (or International Normalized Ratio[INR]) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN or within the intended therapeutic range within 72 hours before the first dose of study drug in subjects receiving anticoagulant therapy
12. Willing and able to comply with scheduled visits, treatment plan, and laboratory tests
13. Absence of any other malignancy which has been active or treated within the past 3 years, except for cervical intraepithelial neoplasia, and nonmelanoma skin cancers (basal cell and squamous cell carcinomas)
14. Men who are sterile (including vasectomy confirmed by post vasectomy semen analysis) OR agree to use a condom with spermicide and to not donate sperm during the study and for at least 90 days following last dose of PT01
15. Female subjects must be postmenopausal (>12 months without menses) or surgically sterile (ie,by hysterectomy and/or bilateral oophorectomy) or must be using highly effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 90 days after their last dose of PT01
16. Subjects who are of childbearing potential must have a negative serum pregnancy test at Screening and within 72 hours prior to the first dose
17. Peripheral forearm veins suitable for venous access including cannulation for infusion of PT01 and multiple blood sampling

Exclusion Criteria:

Eligible subjects must not have/be:

1. Received prior arginase or arginine deiminase therapy
2. Received recent anticancer therapy defined by:

   * Chemotherapy, immunotherapy, hormonal therapy, and monoclonal antibodies (but excluding nitrosourea, mitomycin-C, targeted therapy) ≤28 days prior to starting study drug or who have not recovered from side effects of such therapy to Grade≤1 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v4.03) except for subjects with alopecia; subjects receiving luteinizing hormone-releasing hormone agonists may be considered for enrollment after discussion with the Sponsor
   * Last administration of nitrosourea or mitomycin-C ≤42 days prior to starting study drug or who have not recovered from the side effects of such therapy to Grade ≤1
   * Targeted therapy (eg, sunitinib, sorafenib, pazopanib) ≤14 days prior to starting study drug, or who have not recovered from the side effects of such therapy to Grade ≤1
   * Radiotherapy ≤28 days prior to starting study drug or ≤14 days prior to starting study drug in the case of localized radiotherapy (eg, for analgesic purpose or for lytic lesions at risk of fracture) or who have not recovered from radiotherapy toxicities to Grade ≤1
3. Undergone major surgery (eg, intrathoracic, intraabdominal, or intrapelvic), open biopsy, or significant traumatic injury ≤28 days prior to starting study treatment; subjects who have had minor procedures, percutaneous biopsies, or placement of vascular access device ≤7 days prior to starting study drug; or subjects who have not recovered from side effects of such procedure or injury
4. Uncontrolled concurrent illness including, but not limited to, ongoing or active serious infection Athenex, Inc. Confidential Page 10 Final v2.0_17 Jun 2019 Clinical Study Protocol_Amendment 01 ATX-PT01-001 requiring systemic antimicrobials (within 14 days prior to first dose), uncontrolled arterial hypertension (>160/100 mm Hg on antihypertensive medications), chronic pulmonary disease requiring oxygen, known bleeding disorders, uncontrolled endocrine diseases, altered mental status, or psychiatric illness/social situations that would limit compliance with protocol requirements
5. Significant cardiac or pulmonary disease defined by New York Heart Association Class III or IV, history of myocardial infarction within 6 months prior starting study drug, significant unstable arrhythmia, or evidence of ischemia on ECG
6. Symptomatic or uncontrolled brain metastases requiring current treatment (fewer than 28 days from last cranial radiation or from last steroids use)
7. Healing or open wound(s)
8. Lack of recovery of prior AEs to Grade ≤1 severity (except alopecia or lymphopenia) due to medications administered prior to the first dose of study drug
9. Any other condition or finding (including social situation) that, in the opinion of the Investigator, may render the subject to be either at excessive risk for treatment complications or not able to provide evaluable outcome information
10. Pregnantorbreast-feedingwomen
11. Known allergy to any of the formulation components of PT01

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD), and/or recommended Phase 2 dose (RP2D) together with the biologically effective dose (BED) of PT01. | 4 weeks
  Dose-limiting toxicity (DLT) for determination of MTD and/or RP2D. The grading of toxicity is based on the NCI CTCAE v4.03 criteria.
  Reduction and duration of arginine for determination of BED
Number of participants with treatment-related adverse events as assessed by CTCAE v4.3 criteria. | Day 1 up to 30 days post last dose
  Number of participants with treatment related changes from baseline in vital signs, laboratory parameters and 12-lead ECG findings.

SECONDARY OUTCOMES:
Area Under Plasma Concentration-Time Curve (AUC) | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post dose.
Maximum Observed Plasma Concentration (Cmax) of PT01 | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
The preliminary activity of PT01 by evaluating tumor response. | 8 weeks
  Tumor response according to RECIST v1.1 (best ORR for complete response [CR] and partial response [PR], stable disease, progressive disease), duration of response, PFS Tumor biomarkers in appropriate tumor types
The elimination half-life (t1/2) of PT01 | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
The amount of PT01present at the maximum concentration in plasma (Tmax) | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
The time of last quantifiable presence of PT01 in plasma(Tlast) | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
PT01 concentration at the end of a dosing interval, immediately before next administration (Ctrough), the lowest observed concentration. | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
The volume of PT01 distribution (Vd) in plasma. | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
The total clearance of the PT01 from plasma (CL) | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion
Duration of arginine reduction <10% of baseline. | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion.
The absolute-percent of arginine reduction from baseline | Cycle 0 Day 1: predose PT01 (Hour 0) and at 0.5 (end of infusion), 2, 4, 8, 24, 48, 72, 168, and 240 hours after the start of the PT01 IV infusion. Cycle 1 and Beyond, prepose and .5 hour post infusion

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No